CLINICAL TRIAL: NCT02352259
Title: Treatment of Liver Metastases With Electrochemotherapy (ECTJ) Phase II
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Institute of Oncology Ljubljana (Other)
Collaborators: University Medical Centre Ljubljana (Other); University Medical Centre Maribor (Other); University of Ljubljana (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 03-Z/KESOPKR-28
Record Dates: First submitted 2014-12-17; First posted 2015-02-02 (Estimated); Results first posted 2021-03-24 (Actual); Last update posted 2021-03-24 (Actual); Status verified 2021-03

CONDITIONS: Liver Metastases
Keywords: Liver metastases of colorectal cancer Electrochemotherapy; Bleomycin; Electrochemotherapy
MeSH Terms: interventions — Electrochemotherapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Electrochemotherapy (Experimental)
  Interventions: Procedure: Electrochemotherapy; Device: Cliniporator Vitae®; Drug: Bleomycin PHC 15 e. (United States Pharmacopeia - USP)

INTERVENTIONS:
Procedure: Electrochemotherapy — Treatment procedure: anesthesia, positioning of electrodes, intravenous in bolus administration of bleomycin, within 8-30 min after administration of bleomycin application of electric pulses, removal of electrodes.
Device: Cliniporator Vitae® — Positioning of electrodes, within 8-30 min after administration of bleomycin application of electric pulses (8 pulses, duration 100 microseconds, frequency 4 Hz with amplitude adequate to cover the whole treated lesion with electric field necessary for reversible plasma membrane permeabilization), removal of electrodes.
Drug: Bleomycin PHC 15 e. (United States Pharmacopeia - USP) — Intravenous in bolus administration of bleomycin (15 mg/m2), 8 minutes before application of electric pulses

SUMMARY:
The study is prospective, phase II study, The primary objective of the study is evaluation of the feasibility and safety of intraoperative electrochemotherapy of colorectal liver metastases. The secondary objective is to determine the efficacy of electrochemotherapy treatment, based on histological and radiological evaluation of treated metastases. The endpoints are: toxicity according to the Common Terminology Criteria for Adverse Events (CTCAE) ver. 4.0 and response rate measured by percentage of vital tumor cells and mRECIST criteria.

DETAILED DESCRIPTION:
The study is an extension of previously concluded and published study on electrochemotherapy of colorectal liver metastases (Edhemovic et al. JSO 2014). In this extension 15 patients will be included. Four groups of patients will be included. The patients from groups 1 and 2 are patients with up to 3 unresectable liver metastases, demanding too excessive resection, or untreatable by standard thermal ablative methods due to the close proximity of major blood vessels. Electrochemotherapy will be offered to these patients as the only treatment option. In case of multiple, both resectable and non-resectable liver metastases, the latter will be treated with electrochemotherapy, whereas other metastases will be resected or treated by RFA. These groups of patients are:

1. Patients with one to three (1-3) metachronous liver metastases of colorectal cancer, not larger than 5 cm, that are positioned in unresectable liver area, near blood vessels, but in otherwise operable patients.
2. Recurrent liver metastases of colorectal cancer, not more than 3 and not larger than 5 cm in diameter, each. For those patients any other treatment could represent unacceptable risk due to possibility of insufficient liver residual after resection or less effective radiofrequency ablation due to the proximity of blood vessels.

   Groups 3 and 4 include patients with intent to cure within standard of care using two-stage surgical approach. This two-stage surgical approach will allow adding electrochemotherapy during the first operation and tissue collection for histological analysis during the second operation. Adding electrochemotherapy to these patients will not affect their treatment within standard of care recommended in the current guidelines. These groups of patients are:
3. Patients with synchronous metastases, but their general condition and extent of the disease will not allow simultaneous removal of the primary tumor and metastases. During the first operation, the primary tumor will be removed (colorectal resection) and some of the liver metastases will be treated by electrochemotherapy. About 6 weeks later, during the second operation for liver metastases, both treated and non-treated metastases will be removed with liver resection.
4. Patients with bilateral, multiple, metachronous metastases in whom standard treatment includ two-stage liver resection, due to the extent of the disease and/or their general condition. During the first operation, right portal vein will be ligated and metastases on the left side will be excised or ablated with radiofrequency ablation. At the same time, up to three metastases on the right side were treated with electrochemotherapy. During the second operation, both treated and non-treated metastases on the right side will be removed with right hemihepatectomy.

Electrochemotherapy will be offered to the patients also when they refuse standard treatment.

Depending on the position of metastases, appropriate electrodes will be selected; hexagonal needle electrodes with fixed geometry for metastases not larger than 3 cm in diameter, where their lower edge is located up to 3 cm below the liver capsule. ECT will be performed based on standard operating procedures for treatment of cutaneous and subcutaneous tumors / metastases with ECT.

Individual electrodes, positioned according to the prepared treatment plan will be used for metastases up to 5 cm in diameter, or located near vena cava or large hepatic or portal veins.

Electrochemotherapy will be performed within 8-28 min after intravenous in bolus administration of bleomycin (15 mg/m2).

Triggering of electric pulses will be synchronized with ECG signals, through the ECG triggering device AccuSync to avoid delivery of pulses in vulnerable period of the heart.

All patients will be treated after the procedure has been thoroughly described to them, and have signed informed consent.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically and/or cytologically confirmed colorectal cancer.
2. Age over 18.
3. Life expectancy more than 3 month.
4. Performance status Karnofsky ≥ 70 or (World Health Organization) WHO ≤ 2.
5. Chemotherapy free interval 2-5 weeks, depending on the drugs used.
6. Patient must be mentally capable of understanding the information given.
7. Patient must give informed consent.
8. Patient must be discussed at the multidisciplinary team for tumors of the gastrointestinal tract before entering the trial.

Exclusion Criteria:

1. Secondary primary tumor, except surgically treated noninvasive cancer of cervix, or surgically or irradiated basal cell carcinoma
2. Visceral, bone or diffuse metastases.
3. Life-threatening infection and/or heart failure and/or liver failure and/or other severe systemic pathologies.
4. Clinically significant ascites.
5. Significant reduction in respiratory function.
6. Age less than 18 years.
7. Coagulation disturbances.
8. Cumulative dose of 250 mg/m2 bleomycin received.
9. Allergic reaction to bleomycin.
10. Impaired kidney function (creatinin > 150 µmol/l).
11. Patients with epilepsy.
12. Patients with arrhythmias.
13. Patients with pacemaker or defibrillator.
14. Pregnancy.
15. Patient incapable of understanding the aim of the study or disagree with the entering into the clinical study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 23 (Actual)
Dates: Start 2013-09; Primary Completion 2018-10 (Actual); Study Completion 2018-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gregor Sersa, PhD, Study Director — Institute of Oncology Ljubljana, Ljubljana, Slovenia; Ibrahim Edhemovic, MD, PhD, Principal Investigator — Institute of Oncology Ljubljana, Department of Surgical Oncology, Ljubljana, Slovenia
Locations (4):
- Slovenia (4):
  - Faculty of Electrical Engineering, University of Ljubljana, Slovenia, Ljubljana
  - Institute of Oncology Ljubljana, Ljubljana
  - University Medical Centre Ljubljana, Ljubljana, Slovenia, Ljubljana
  - University Medical Centre Maribor, Maribor, Slovenia, Maribor

REFERENCES:
- [Background] Edhemovic I, Brecelj E, Gasljevic G, Marolt Music M, Gorjup V, Mali B, Jarm T, Kos B, Pavliha D, Grcar Kuzmanov B, Cemazar M, Snoj M, Miklavcic D, Gadzijev EM, Sersa G. Intraoperative electrochemotherapy of colorectal liver metastases. J Surg Oncol. 2014 Sep;110(3):320-7. doi: 10.1002/jso.23625. Epub 2014 Apr 30. PMID 24782355
- [Background] Edhemovic I, Gadzijev EM, Brecelj E, Miklavcic D, Kos B, Zupanic A, Mali B, Jarm T, Pavliha D, Marcan M, Gasljevic G, Gorjup V, Music M, Vavpotic TP, Cemazar M, Snoj M, Sersa G. Electrochemotherapy: a new technological approach in treatment of metastases in the liver. Technol Cancer Res Treat. 2011 Oct;10(5):475-85. doi: 10.7785/tcrt.2012.500224. PMID 21895032

RESULTS

PARTICIPANT FLOW:
Groups:
- Electrochemotherapy: All patients were administered with intravenous bolus of bleomycin (15,000 IU/m2, Bleomycin medac, Medac, Hamburg, Germany), after intraoperative ultrasound confirmed the correct electrode placement. Eight minutes after bleomycin injection, electric pulses were delivered by Cliniporator®VITAE (IGEA SpA, Carpi, Italy).
Period: Overall Study
Arm/Group | Electrochemotherapy
Started | 23
Completed | 23
Not Completed | 0

BASELINE CHARACTERISTICS:
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 9
  >=65 years | 14
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 17
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 23
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Number; unit: participants]
  Slovenia | 23
CRC liver metastases [Number; unit: metastases] — Patients presented with CRC liver metastases
  metastases | 23

OUTCOME MEASURES:

1. Primary Outcome: Evaluation of Safety Related to Electrochemotherapy
Description: Recording of adverse events according to CTCAE criteria
Time Frame: After operation on day 7
Measure: Count of Participants; unit: Participants
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 23
Participants
  No adverse events | 20
  ECT nonrelated mild adverse avents | 3
  ECT related mild adverse avents | 0
  Adverse avents | 0

2. Secondary Outcome: Response to Treatment (Determined by Modified RECIST Criteria).
Description: Response Evaluation Criteria In Solid Tumors Criteria (RECIST v1.0) for target lesions and assessed by MRI/CT:
  Complete Response (CR), Disappearance of all target lesions; Partial Response (PR), >=30% decrease in the sum of the longest diameter of target lesions; Overall Response (OR) = CR + PR
Time Frame: After operation on the days 30, 60, 90 and 120
Measure: Count of Participants; unit: Participants
Arm/Group | Electrochemotherapy
Number analyzed (Participants) | 23
Participants
  complete response (CR) | 10
  partial response (PR) | 4
  progressive disease (PD) | 9

ADVERSE EVENTS:
Time Frame: 7, 30, 60, 90, 120 days
Description: adverse events observed in 3 out of 23 patients, no serious adverse events
Arm/Group | Electrochemotherapy
All-Cause Mortality (participants affected / at risk) | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23
Other Adverse Events (participants affected / at risk) | 3/23
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Electrochemotherapy (N=23)
SIRS (Infections and infestations) | 1 — Systemic inflammatory response syndrome
arrhythmia (Cardiac disorders) | 1 — arrhythmia
abscess (Hepatobiliary disorders) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Informed Consent Form (2013-03-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT02352259/ICF_000.pdf
  • Study Protocol and Statistical Analysis Plan (2013-03-30): https://cdn.clinicaltrials.gov/large-docs/59/NCT02352259/Prot_SAP_001.pdf